CLINICAL TRIAL: NCT03869918
Title: Comparative Effectiveness of Integrated Exercise and Urge Suppression Verses Usual Care for Reducing the Risk of Falls in Women With Urgency Urinary Incontinence
Brief Title: Physical Exercise and Bladder Training Program for Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 819469
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: A pilot randomized comparative effectiveness trial of integrated exercise and urge suppression versus usual care in older women with UUI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Participant is assigned to undergo standard of care.
- Exercise Group (Experimental): If the participant is assigned to the exercise group, she will either exercise at home or take a class at the participating facility under the supervision of an instructor.
  Interventions: Other: Exercise Program
- Observational Group (No Intervention): If a subject is eligible, but does not want to exercise, she will be in a third group that is an observation group.

INTERVENTIONS:
Other: Exercise Program — Exercise at home or through a class as chosen by the subject.
  Arms: Exercise Group

SUMMARY:
The overall objective of this project is to reduce the risk of falls in elderly community dwelling women over 60 years of age with urgency urinary incontinence (UUI). In this pilot study, the investigators plan to develop, validate and test a home based integrated exercise and urge suppression intervention (bladder training) that targets functional mobility, reduces anxiety urgency and physical barriers and is implemented in partnership with all stakeholders. Key eligibility criteria: women over 60 years of age, with moderate to severe UUI, and low physical activity.

DETAILED DESCRIPTION:
Over 40% women age 65 and older or an estimated million women in the US suffer from urgency urinary incontinence (UUI), a condition characterized by urgency to urinate. UUI is a well-known marker for frailty and older women with UUI are at two fold higher risk for falls. According to the biopsycho- ecological paradigm, UUI and its associated falls are the result of interaction of the patients physical abilities (bladder urgency and reduced balance and strength to reach the toilet), mental attitudes (anxiety related to urgency, shame and stigma of leakage), social expectations (life demand and roles that limit access to bathroom), and physical environment (physical barriers to reach the toilet).

Anti-muscarinic medications, the most common treatment for UUI, address only bladder urgency and their side-effects may exacerbate falls. The investigators plan an innovative treatment approach that will integrate each of the bio-psycho-ecological levels implicated in UUI and falls. Strength and balance exercises improve functional mobility and have been shown to reduce both fall risk as well as UUI in high risk frail older adults. Behavioral urge suppression reduces anxiety related to urgency and improves mental abilities to handle life demands and roles. Simple home improvements can reduce environmental barriers. Adherence is an important barrier in the implementation of exercise and behavior modification. Prior studies, including those by the investigators, have shown that preferred treatments are associated with improved adherence, satisfaction and outcomes in women with UUI. The investigators hypothesize that an integrated exercise and urge suppression program targeted to improving physical performance relevant to continence behavior will reduce the risk of falls in appropriately selected community dwelling women with urinary incontinence. In this pilot study, the investigators plan to develop, validate and test a home based integrated exercise and urge suppression intervention that targets functional mobility, reduces anxiety urgency and physical barriers and is implemented in partnership with all stakeholders. The proposed pilot study for a planned submission in June 2014 fulfills PCORIs national priorities and research agenda through improving patient centered outcome measures, informed decision making based on risks and benefits, innovative Page 9 of 17 community based delivery of the intervention, addressing barriers to care, and engaging all stakeholders involved in the care of older women with UUI including patients, providers, and community advocates.

The overall objective of this project is to reduce the risk of falls in elderly frail community dwelling women with urgency urinary incontinence (UUI). The specific aim is: To determine the feasibility of enrollment and randomization of a comparative effectiveness trial of integrated exercise and urge suppression program versus usual care in older community dwelling women with urge urinary incontinence. Hypothesis: Older women with UUI who receive their preferred treatment option, exercises and urge suppression, will have better objective (fewer functional limitations, falls risk and urinary incontinence) and subjective (HRQOL, satisfaction with care, and psychological wellbeing) outcomes than women who receive usual care.

ELIGIBILITY:
Inclusion Criteria:

1. female
2. age 60+ years
3. community dwelling
4. Moderate to severe UUI (as measured by International Consultation on Incontinence Questionnaire Short Form)
5. low physical activity (Physical Activity Staging questionnaire)
6. cognitively able to complete the study (in opinion of the referring provider) Women currently on anti-cholinergic medication for urinary incontinence will be allowed if particpants meet the above criteria.

Exclusion Criteria:

1. cognitive impairment (in opinion of the referring provider)
2. unable to provide informed consent or communicate in English
3. desire for surgical management
4. osteoporosis
5. lack of medical clearance from the physician.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-03-30 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Physical Function as measured by the Short Physical Performance Battery | 2 months
  An objective measure of physical function as measured by the Short Physical Performance Battery that measures balance, gait speed, and lower extremity strength and has high validity and sensitivity to change for predicting fall risk.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No